CLINICAL TRIAL: NCT05542797
Title: Comparison of Dydrogesterone and Micronized Progesterone Treatments in the Treatment of Threatened Miscarriage.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Hasan Ali Inal, MD, obstetrics and gynecology, Konya Meram State Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 351508
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Miscarriage Threatening
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micronised progesterone (Experimental): Micronized progesterone will be given to 70 pregnant women with threated miscarriage.
  Interventions: Drug: Duphastone
- Dydrogesterone (Experimental): Dydrogesterone will be given to 70 pregnant women with threated miscarriage.
  Interventions: Drug: Duphastone

INTERVENTIONS:
Drug: Duphastone — dydrogesterone hormone

SUMMARY:
In this study, we aimed to compare the effects of two drugs used for the threated miscarriage on the miscarriage rate.

DETAILED DESCRIPTION:
About 140 pregnant women who applied to our clinic due to the threated miscarriage in the first trimester will be randomly given micronized progesterone to half and dydrogesterone to the other half. After the treatment, the miscarriage rates in the groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with threated miscarriage in the first trimester.

Exclusion Criteria:

* - pregnant women with abortus incipiens.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Miscarriage rate | One year
  Effects of two drugs to be used on live birth rate in pregnant women with threated miscarriage

IPD SHARING:
Plan to Share IPD: No